CLINICAL TRIAL: NCT06157801
Title: Evaluation of Hereditary Cancer Educational Videos
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0654; NCI-2023-10074 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Hereditary Cancer
MeSH Terms: interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interview Study: In the interview study, participants will watch the video, then complete an interview. This will take about 50 minutes.
  Interventions: Behavioral: Interview Study
- Survey Study: In the survey study, participants will complete a survey about your education and complete a quick test about your knowledge of hereditary cancer. Participants will then watch the video. complete another survey similar to the one before the video. This should take about 30 minutes.
  Interventions: Behavioral: Survey Study

INTERVENTIONS:
Behavioral: Interview Study — All study participants will have the following demographic information collected from their medical records:
  * Sex (Male/Female/Other)
  * Date of birth
  * Preferred language (English/Spanish)
  * Health insurance status (for example: private insurance, HCHD "gold card")
  * Cancer diagnosis (if yes: cancer type/organ, date of pathology diagnosis)
  * Genetic testing result (gene with pathogenic/likely pathogenic variant)
  * Date of genetic testing result
  * Date of documented result disclosure.
  Groups: Interview Study
Behavioral: Survey Study — All study participants will have the following demographic information collected from their medical records:
  * Sex (Male/Female/Other)
  * Date of birth
  * Preferred language (English/Spanish)
  * Health insurance status (for example: private insurance, HCHD "gold card")
  * Cancer diagnosis (if yes: cancer type/organ, date of pathology diagnosis)
  * Genetic testing result (gene with pathogenic/likely pathogenic variant)
  * Date of genetic testing result
  * Date of documented result disclosure.
  Groups: Survey Study

SUMMARY:
To learn if educational videos can help participants be more informed about hereditary cancers (ones that run in the family).

DETAILED DESCRIPTION:
Primary Objective

Determine the impact of educational videos on:

* Participant's hereditary cancer knowledge.
* Participant's confidence to share hereditary cancer information with family members.

Secondary Objective

* Determine impact of educational videos on participant's confidence to undergo hereditary cancer screening.
* Identify opportunities to tailor and improve the educational video's content, style, and understandability per participant preferences and feedback.

ELIGIBILITY:
Inclusion Criteria:

1. Participants of The Harris Health System Lyndon B. Johnson (LBJ) Hospital outpatient oncology clinics (i.e., Gynecologic Oncology, Medical Oncology).
2. 18 years of age or older.
3. Speaks and/or reads English or Spanish.
4. Has a pathogenic or likely pathogenic variant (mutation) in BRCA1, BRCA2, MLH1, MSH2, MSH6, PMS2, and/or EPCAM on germline genetic testing.
5. Has a documented genetic testing results disclosure encounter (i.e. telephone call, follow-up appointment).

Exclusion Criteria:

1. No longer receives outpatient care at LBJ Hospital at time of recruitment.
2. Has only a variant of uncertain significance in BRCA1, BRCA2, MLH1, MSH2, MSH6, PMS2, and/or EPCAM.
3. Has only a pathogenic or likely pathogenic variant in gene other than BRCA1, BRCA2, MLH1, MSH2, MSH6, PMS2, or EPCAM.
4. Is unwilling, unable, or requires a legally authorized representative to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Harris Health System (LBJ Hospital)
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Hereditary Cancer Multidimensional Measure of Informed Choice Questionnaires | through study completion; an average of 1 year
  Hereditary Cancer Multidimensional Measure of Informed Choice (MMIC)
  Knowledge Score scale: (1-8) true or false

CONTACTS AND LOCATIONS:
Overall Officials: Jose Rauh-Hain, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org